CLINICAL TRIAL: NCT07198724
Title: ERADICATE: A Phase Ib/II Study of Elacestrant Plus Trastuzumab Deruxtecan in Patients With CDK4/6 Inhibitor and Endocrine-resistant HR+/HER2-low or HER2-ultralow Metastatic Breast Cancer
Acronym: ERADICATE
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sarah Sammons, MD (Other)
Collaborators: Stemline Therapeutics, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Sarah Sammons, MD, Sponsor-Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 25-437
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Breast Cancer; HER2 Low Breast Carcinoma; HER2-negative Breast Cancer; Breast Cancer; Breast Cancer Female
Keywords: Metastatic Breast Cancer; HER2 Low Breast Carcinoma; HER2-negative Breast Cancer; Breast Cancer; Breast Cancer Female; HR+/HER2-low Breast Cancer; HR+/HER2-ultralow Breast Cancer; Endocrine-resistant Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — elacestrant; RAD1901; trastuzumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1b: Elacestrant + Trastuzumab Deruxtecan (Experimental): Up to 28 participants will be enrolled to determine the recommended phase 2 dosage of Elacestrant and will complete the following:
  * Baseline visit
  * Cycle 1 (21 day cycle)
    * Days 1 through 21: Predetermined dose of Elacestrant 1x daily.
    * Day 1: Predetermined dose of Trastuzumab Deruxtecan 1x daily.
  * Cycle 2 through End of Treatment (21 day cycle):
    * Imaging every 9 weeks until Cycle 9, then every 12 weeks
    * Day 1: tumor biopsy
    * Days 1 through 21: Predetermined dose of Elacestrant 1x daily.
    * Day 1: Predetermined dose of Trastuzumab Deruxtecan 1x daily.
    * End of Treatment visit with imaging
    * Follow up visits every 6 months
    * If 3 or less out of 12 participants experience a dose-limiting toxicity (DLT), the recommended Phase II dose of Elacestrant will be that dose level. If there are 4 or more DLTs, Elacestrant dosage will de-escalate and 12 more participants will be enrolled.
  Interventions: Drug: Elacestrant; Drug: Trastuzumab Deruxtecan
- Phase 2: Elacestrant + Trastuzumab Deruxtecan (Experimental): 37 participants will complete the following:
  * Baseline visit
    -Cycle 1 (21 day cycle)
  * Days 1 through 21: Predetermined dose of Elacestrant 1x daily.
  * Day 1: Predetermined dose of Trastuzumab Deruxtecan 1x daily.
    -Cycle 2 through End of Treatment (21 day cycle):
  * Imaging every 9 weeks until Cycle 9, then every 12 weeks
  * Day 1: tumor biopsy
  * Days 1 through 21: Predetermined dose of Elacestrant 1x daily.
  * Day 1: Predetermined dose of Trastuzumab Deruxtecan 1x daily.
  * End of Treatment visit with imaging
  * Follow up visits every 6 months
  Interventions: Drug: Elacestrant; Drug: Trastuzumab Deruxtecan

INTERVENTIONS:
Drug: Elacestrant — Selective estrogen receptor degrader (SERD), film-coated tablet, taken orally per protocol.
  Other Names: Elacestrant dihydrochloride; RAD1901
Drug: Trastuzumab Deruxtecan — HER2-directed antibody-drug conjugate, vial, via intravenous (into the vein) infusion per standard of care
  Other Names: Fam-Trastuzumab; ENHERTU; DS-8201a; T-DXd

SUMMARY:
The goal of this study is to evaluate the safety and efficacy of elacestrant in combination with trastuzumab deruxtecan (T-DXd) in participants with hormone receptor-positive (HR+), HER2-low or HER2-ultralow, metastatic breast cancer that is resistant to prior CDK4/6 inhibitor and endocrine therapy.

The names of the study drugs involved in this study are:

* Elacestrant (a type of selective estrogen receptor degrader)
* Trastuzumab deruxtecan (a type of standard of care antibody drug conjugate)

DETAILED DESCRIPTION:
This phase Ib/II, open-label, single-arm, investigator-initiated study is to evaluate the safety and efficacy of elacestrant in combination with trastuzumab deruxtecan (T-DXd) in participants with hormone receptor-positive (HR+), HER2-low or HER2-ultralow, metastatic breast cancer that is resistant to prior CDK4/6 inhibitor and endocrine therapy.

This is a Phase I/II clinical trial. A Phase I clinical trial tests the safety of an investigational drug and also tries to define the appropriate dose of the investigational dose to use for further studies. "Investigational" means that the drug is being studied.

The phase Ib dose-escalation portion of the study is to determine the recommended phase II dose (RP2D) of the Elacestrant in combination with trastuzumab deruxtecan, followed by a phase II expansion to further evaluate efficacy and safety at the RP2D.

The research study procedures include screening for eligibility, in-clinic visits, blood tests, urine tests, Computerized Tomography (CT) scans, Magnetic Resonance Imaging (MRI) scans, electrocardiograms (ECGs), and tumor biopsies.

The U.S. Food and Drug Administration (FDA) has not approved Elacestrant for CDK4/6 inhibitor and endocrine-resistant HR+/HER2-low or HER2-ultralow metastatic breast cancer but it has been approved for ER-positive, HER2-negative, ESR1-mutated advanced or metastatic breast cancer.

The FDA has approved trastuzumab deruxtecan as a treatment option for CDK4/6 inhibitor and endocrine-resistant HR+/HER2-low or HER2-ultralow metastatic breast cancer.

The FDA has not approved the combination of Elacestrant and Trastuzumab deruxtecan for CDK4/6 inhibitor and endocrine-resistant HR+/HER2-low or HER2-ultralow metastatic breast cancer.

It is expected that about 65 people will take part in this research study.

Stemline-Menarini is supporting this research study by providing the study drug, Elacestrant.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a histologically or cytologically confirmed diagnosis of HR+/HER2-low metastatic or unresectable locally advanced breast cancer, defined as ER ≥ 10%, any PR in the most recent sample and HER2-low (IHC 1+ or IHC 2+ and ISH non-amplified) or HER2-ultralow (IHC 0 and any membranous staining on any prior sample). Cutoff values for positive/negative HER2 staining should be in accordance with current ASCO/CAP (American Society of Clinical Oncology/College of American Pathologists) guidelines.76 Participants without pathologic or cytologic confirmation of metastatic disease should have unequivocal evidence of metastasis from physical examination or radiographic evaluation.
* Participants must have had prior CDK4/6 inhibitor and either:

  * Disease progression on or within 12 months of endocrine therapy plus a CDK4/6 inhibitor in the adjuvant setting
  * One previous line of endocrine therapy in metastatic setting if disease progression within 6 months of first-line CDK4/6 plus endocrine treatment for metastatic disease or disease recurrence within 24 months after initiation of adjuvant endocrine therapy
  * Two previous lines of endocrine therapy in the metastatic with or without a targeted therapy (such as but not limited to CDK4/6, mTOR, or PI3K inhibitors) administered for the treatment of metastatic disease.
  * Of note with regards to the 2 lines of previous endocrine therapy requirement:- Disease recurrence while on the first 24 months of adjuvant endocrine therapy will be considered a line of therapy; these patients will only require 1 line of endocrine therapy in the metastatic setting.

    * Single-agent PARP inhibitor therapy is not considered a line of endocrine therapy but is allowed.
    * Changes in dosing schedules, or discontinuations/restarting of the same drugs of the addition of a targeted therapy to an endocrine therapy without progression (e.g., adding a CDK4/6 inhibitor to a current aromatase inhibitor regimen) will not be considered separate lines of therapy.
* Participants may have not received prior chemotherapy or ADC in the metastatic setting.
* Participants must have measurable disease per RECIST 1.1 criteria. See Section 11 for the definition of measurable disease. Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm (≥2 cm) by chest x-ray or as ≥10 mm (≥1 cm) with CT scan, MRI, or calipers by clinical exam. See Section 12 (Measurement of Effect) for the evaluation of measurable disease.
* Participants must have known ESR1 mutation status in tumor or ctDNA within 6 months of enrollment to the trial.
* Women or men age ≥18 years are eligible.
* ECOG performance status ≤ 2.
* Participants must meet the following organ and marrow function as defined below:

  * Absolute neutrophil count ≥ 1,500/µL
  * Platelets ≥ 100,000/µL
  * Hemoglobin ≥ 9.0 g/dL
  * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) (or ≤ 2 x ULN in patients with documented Gilbert's syndrome)
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 x institutional ULN (or < 5 x ULN in patients with liver metastases)
  * Creatinine ≤ 1.5 x institutional ULN OR
  * Calculated creatinine clearance ≥ 45 mL/min via the Cockcroft-Gault formula for participants with creatinine levels above institutional ULN
  * Participants with a history of central nervous system (CNS) metastases are eligible if: Stable or untreated, asymptomatic brain metastases not needing immediate local therapy. For patients with untreated CNS lesions > 2.0 cm on screening contrast brain MRI, discussion with and approval from the medical monitor is required prior to enrollment.
  * Previously treated brain metastases

    * a. Brain metastases previously treated with local therapy may either be stable since treatment or may have progressed since prior local CNS therapy, provided that there is no clinical indication for immediate re-treatment with local therapy in the opinion of the investigator
    * b. Patients treated with CNS local therapy for newly identified lesions may be eligible to enroll if all of the following criteria are met: i. Time since WBRT is ≥ 14 days prior to first dose of treatment, time since SRS is ≥ 7 days prior to first dose of treatment, or time since surgical resection is ≥ 14 days
* Women must be postmenopausal, which is defined as any of the following:

  * Age ≥ 60 years
  * Age < 60 and amenorrhea for 12 or more months (in the absence of chemotherapy, tamoxifen, toremifene, or ovarian suppression) and FSH, and estradiol in the postmenopausal range per local normal range
  * Premenopausal women must be on GnRH agonist prior to study entry are eligible. Women in this group MUST remain on the GnRH agonist for the duration of protocol treatment.
  * Status-post bilateral oophorectomy - After adequate healing post-surgery
* Premenopausal women must have a negative serum or urine pregnancy test. Pregnancy testing does not need to be pursued in female participants who are:

  * Age > 60 years; or
  * Age < 60 with intact uterus and amenorrhea for 12 consecutive months or more AND estrogen (estradiol) levels within postmenopausal range; or
  * Status-post bilateral oophorectomy, total hysterectomy, or bilateral tubal ligation
* The effects of elacestrant and T-DXd on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Women treated or enrolled on this protocol must use an effective method of birth control for 4 months after the last dose of elacestrant or 7 months after the last dose of trastuzumab deruxtecan, whichever is later. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of elacestrant and T-DXd administration.

  * Adequate contraception is defined as one highly effective non-hormonal form of contraception or two effective forms of non-hormonal contraception by the participant and/or partner.
  * Highly Effective Non-Hormonal Contraception Methods of birth control which result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly are considered highly effective forms of contraception.
  * The following non-hormonal methods of contraception are acceptable:

    * True abstinence when this is in line with the preferred and usual lifestyle of the participant. [Periodic abstinence (e.g., calendar, ovulation, symptothermal post- ovulation methods) and withdrawal are not acceptable methods of contraception].
    * Male sterilization (with appropriate post-vasectomy documentation of the absence of sperm in the ejaculate). For female participants, the vasectomized male partner should be the sole partner.
* Participants must be able to swallow and retain oral medication.
* Participants must be willing to undergo two mandatory research biopsies (one at baseline, one during treatment) if tumor is safely accessible.
* Ability to understand and the willingness to sign a written informed consent document. (Providing consents in as many languages as possible is encouraged)

Exclusion Criteria:

* Prior treatment with an antibody-drug conjugate in any setting.
* Prior treatment with an oral novel estrogen receptor degrader or modulator in the metastatic setting (SERD, SERM, PROTAC, or CERAN). Prior fulvestrant is allowed. A washout period of 7 days is required for any endocrine or targeted therapy.
* Patients with known brain metastases that are symptomatic or that require therapy for symptom control are not eligible. Patients with stable or asymptomatic brain metastases are allowed. Participants with CNS metastases treated by neurosurgical resection or brain biopsy performed within 4 weeks before day 1 of study therapy will be excluded.
* Receipt of any other investigational compound or device within 2 weeks of the first dose of treatment in this study.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to elacestrant or T-DXd.
* History of (non-infectious) pneumonitis that required steroids or current ILD by imaging at screening.
* Patients who are pregnant or breastfeeding, or who expect to become pregnant within the projected duration of the study (starting with the screening visit through 12 months after the last dose of study treatment for participants who have received cyclophosphamide, and for 6 months after the last dose of study treatment for those who have not).
* Patients with a known history of active tuberculosis.
* Uncontrolled intercurrent illness including, but not limited to: ongoing or active infection requiring systemic therapy, clinically significant cardiovascular disease including: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication, uncontrolled diabetes mellitus, gastrointestinal disorders potentially affecting the absorption of elacestrant, inflammatory bowel disease or chronic diarrhea, short bowel syndrome, or total gastric resection, or psychiatric illness/social situations that would limit compliance with study requirements. Active hepatitis B or active hepatitis C infection. Ability to comply with study requirements is to be assessed by each investigator at the time of screening for study participation.
* Patients with a history of different malignancy are ineligible, except for those who have been disease-free for at least three years and are deemed by the investigator to be at low risk for recurrence of the prior malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: ductal carcinoma in situ of the breast, cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin.
* Significant cardiovascular disease, such as: history of myocardial infarction, acute coronary syndrome or coronary angioplasty/stenting/bypass grafting within the last six months OR congestive heart failure (CHF) New York Heart Association (NYHA) Class II-IV or history of CHF NYHA Class III or IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2038-06-01 (Estimated)

PRIMARY OUTCOMES:
Recommended phase II dose (RP2D) | Assessed at the end of the first treatment cycle, Day 21.
  The RP2D is defined as the dose at which ≤ 3 out of 12 participants experience Dose Limiting Toxicities (DLT) during the first treatment cycle.
Objective Response Rate (ORR) | assessed for response every 9 weeks (3 cycles) +/- 7 days for the first 27 weeks, then every 12 weeks +/- 7 days, and at end of treatment or start of new anticancer therapy, or up to approximately 24 months
  ORR per RECIST 1.1 is defined as the percentage of participants with confirmed complete or partial response as the best overall response.

SECONDARY OUTCOMES:
ORR in Participants with ESR1-mutant endocrine- and CDK4/6 inhibitor-resistant HR+/HER2-low or HER2-ultralow metastatic breast cancer | assessed for response every 9 weeks (3 cycles) +/- 7 days for the first 27 weeks, then every 12 weeks +/- 7 days, and at end of treatment or start of new anticancer therapy, or up to approximately 24 months
  ORR per RECIST 1.1 is defined as the percentage of participants with confirmed complete or partial response as the best overall response.
Clinical Benefit Rate (CBR) | assessed for response every 9 weeks (3 cycles) +/- 7 days for the first 27 weeks, then every 12 weeks +/- 7 days, and at end of treatment or start of new anticancer therapy, or up to approximately 24 months
  CBR per RECIST 1.1 is defined as the percentage of participants with confirmed complete or partial response, or stable disease for ≥ 24 weeks as the best overall response
CBR in Participants with ESR1-mutant endocrine- and CDK 4/6 inhibitor-resistant HR+/HER2-low of HER2-ultralow metastatic cancer | assessed for response every 9 weeks (3 cycles) +/- 7 days for the first 27 weeks, then every 12 weeks +/- 7 days, and at end of treatment or start of new anticancer therapy, or up to approximately 24 months
  CBR per RECIST 1.1 is defined as the percentage of participants with confirmed complete or partial response, or stable disease for ≥ 24 weeks as the best overall response
Median progression-free survival (PFS) | assessed for response/progression every 9 weeks (3 cycles) +/- 7 days for the first 27 weeks, then every 12 weeks +/- 7 days, and at end of treatment or start of new anticancer therapy, or up to approximately 36 months
  PFS is defined as the time from registration to the earlier of progression or death due to any cause. Participants alive without disease progression are censored at date of last disease evaluation.
Median PFS in Participants with ESR1-mutant endocrine- and CDK4/6 inhibitor-resistant HR+/HER2-low or HER2-ultralow metastatic breast cancer | assessed for response/progression every 9 weeks (3 cycles) +/- 7 days for the first 27 weeks, then every 12 weeks +/- 7 days, and at end of treatment or start of new anticancer therapy, or up to approximately 36 months
  PFS is defined as the time from registration to the earlier of progression or death due to any cause. Participants alive without disease progression are censored at date of last disease evaluation.
Median Overall Survival (OS) | assessed at all study visits; once progression is documented, subjects will be followed for survival every 6 months from the time of documented progression until participant withdrawal, death, or removal from study, or up to approximately 36 months
  OS is defined as the time from registration to death due to any cause. Participants still living are censored at the date last known alive.
Median OS in Participants with ESR1-mutant endocrine- and CDK4/6 inhibitor-resistant HR+/HER2-low or HER2-ultralow metastatic breast cancer | assessed at all study visits; once progression is documented, subjects will be followed for survival every 6 months from the time of documented progression until participant withdrawal, death, or removal from study, or up to approximately 36 months
  OS is defined as the time from registration to death due to any cause. Participants still living are censored at the date last known alive.
Duration of Response (DOR) | assessed for response/progression every 9 weeks (3 cycles) +/- 7 days for the first 27 weeks, then every 12 weeks +/- 7 days, and at end of treatment or start of new anticancer therapy, or up to approximately 36 months
  DOR is defined as the time when measurement criteria are met for confirmed complete or partial response (whichever is first recorded) to the first date that recurrent or progressive disease is objectively documented. Participants without response reported are censored at the last disease evaluation.
DOR in Participants with ESR1-mutant endocrine- and CDK4/6 inhibitor-resistant HR+/HER2-low or HER2-ultralow metastatic breast cancer | assessed for response/progression every 9 weeks (3 cycles) +/- 7 days for the first 27 weeks, then every 12 weeks +/- 7 days, and at end of treatment or start of new anticancer therapy, or up to approximately 36 months
  DOR is defined as the time when measurement criteria are met for confirmed complete or partial response (whichever is first recorded) to the first date that recurrent or progressive disease is objectively documented. Participants without response reported are censored at the last disease evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Sammons, MD, Study Director — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu